CLINICAL TRIAL: NCT06142747
Title: SUper-Resolution Ultrasound Imaging of Erythrocytes (SURE) in Normal and Tendinopathic Tendons
Brief Title: Tracking of Red Blood Cells Using Super Resolution Ultrasound in Persons With Healthy or Overuse Injured Tendons
Acronym: SURE-TEND
Status: Recruiting | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: Technical University of Denmark (Other)
Responsible Party: Principal Investigator, René B. Svensson, Senior Researcher, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: BBH161; 854796 (Other Grant/Funding Number: European Research Council: Synergy Grant)
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Tendinopathy
Keywords: Tendon Overuse Injury; Achilles Tendon; Patellar Tendon; Ultrasonography
MeSH Terms: conditions — Tendinopathy | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (3):
- Control: Healthy Controls. Super-Resolution Ultrasound Imaging of Erythrocytes (SURE) of both Achilles and Patellar Tendons.
  Interventions: Diagnostic Test: Super-Resolution Ultrasound Imaging of Erythrocytes (SURE)
- Tendinopathy Achilles: Patients with Achilles Tendinopathy. Super-Resolution Ultrasound Imaging of Erythrocytes (SURE) of Achilles Tendons.
  Interventions: Diagnostic Test: Super-Resolution Ultrasound Imaging of Erythrocytes (SURE)
- Tendinopathy Patellar: Patients with Patellar Tendinopathy. Super-Resolution Ultrasound Imaging of Erythrocytes (SURE) of Patellar Tendons.
  Interventions: Diagnostic Test: Super-Resolution Ultrasound Imaging of Erythrocytes (SURE)

INTERVENTIONS:
Diagnostic Test: Super-Resolution Ultrasound Imaging of Erythrocytes (SURE) — Research ultrasound sequence for tracking erythrocytes and thereby generating a super-resolution image of the vasculature.
  Other Names: Ultrasonography

SUMMARY:
The goal of this observational study is to test whether a new ultrasound method, called SUper Resolution ultrasound imaging of Erythrocytes (SURE), can image the small blood vessels found in tendons of persons with a tendon overuse injury (tendinopathy). The main questions it aims to answer are:

* Is the method sensitive enough to detect the smallest blood vessels
* What information about the blood flow can be obtained (flow velocity, pressure, shape of the vessels)
* Can the flow in an injured tendon be distinguished from that of a healthy one

Participants will receive a non-invasive ultrasound examination of their Achilles (heel) or patellar (knee) tendon, using an advanced high frequency research ultrasound system.

Researchers will compare participants with either an Achilles or patellar tendon overuse injury to participants with healthy tendons, to see if there are distinct differences in the blood vessels that could help diagnose and treat the injuries.

DETAILED DESCRIPTION:
Studies have reported an enlargement of the microvascular network in human tendons with a chronic overuse injury (tendinopathy). Ingrowth of new vessels and accompanying nerves have been proposed to be the cause of painful symptoms in patients with tendinopathy. Doppler ultrasound is the most common imaging modality to clinically investigate tendon neovascularization. This measurement is clinically useful, but its sensitivity is limited, which means that no Doppler flow is visible in healthy tendons despite invasive techniques having shown the presence of such flow. The lack of sensitivity in Doppler ultrasound means that it is impossible to accurately follow the progression from the healthy state (with zero Doppler) to a chronic state (with detectable Doppler), as well as the reverse process during healing of the injury.

The present study is designed to evaluate an ultrasound method called Super-resolution ultrasound imaging of erythrocytes (SURE), which is a new imaging technique for visualization and quantification of the microvasculature of tissues. The method is built on a technique called super-resolution ultrasound imaging (SRI), where an ultrasound contrast agent is injected into the bloodstream and tracked inside the vessels to build an image of the microvasculature. With SURE, no contrast agent is needed; it relies only on standard ultrasound to track the erythrocytes and thereby avoid invasive procedures.

The aim of this study is to determine the applicability of the SURE technique to detecting microvascular flow changes with tendinopathy by quantifying flow parameters in SURE images of healthy and tendinopathic tissues.

The study is designed as a cross-sectional, single-center, diagnostic, case-control trial on participants who are either healthy or have had a tendinopathy in their Achilles or patellar tendon. A formal sample size estimate cannot be made since the SURE method has not been clinically applied before, the sample sizes are therefore based on our experience with other outcomes for this patient group.

The study-specific medical device consists of 2 main components: a scanner system and an ultrasound probe.

* The ultrasound scanner: Vantage 256™ scanner (Verasonics, Kirkland, Washington, USA).
* The probe: Either a GE L8-18i-D linear transducer (GE Healthcare, Chicago, Illinois, USA), or a Vermon RC6gV row-column transducer (Vermon, Tours, France).

Both components are marked for conformity within the European Union (CE). The entire system (including the probe and scanner system) would classify as a Class IIa medical device, but it has not gone through a notified body as the system is not intended for commercial use.

For measurements, the participant is placed on a bed and scanned with conventional ultrasound to locate the region of tendon injury (or the thickest part of the tendon for healthy participants) and characterize it with grey-scale and Doppler imaging. The region of interest is marked on the skin and the ultrasound probe is affixed to the tendon at the specified location using a custom holder to minimize motion. The probe is then be disconnected from the conventional ultrasound scanner and connected to the Vantage 256™ scanner to record SURE images. Image data may be collected for up to 1 minute. Two scans at the same location are used for estimating repeatability. The imaging setup and image processing will be adjusted to maximize quality of the SURE images. From the images, the vessel density, and potentially other parameters (flow rate, flow orientation, vessel dimensions etc.) may be determined.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years of age.
* BMI below 30.
* Able to lie still for 1 minute.
* Capable of providing signed informed consent.

Exclusion Criteria:

* Pregnancy.
* Dementia.
* Smoking.
* Diabetes.
* Arthritis.
* Current or historical injuries to the tendon or surrounding tissue aside from tendinopathy.
* Medical or surgical treatments for their tendinopathy that may influence blood flow.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy participants:
  Persons who have no self-reported current or historical injuries to the tendon and surrounding tissue, and display no symptoms of tendinopathy upon examination.
  Participants with tendinopathy:
  Persons who have no self-reported current or historical injuries to the tendon and surrounding tissue, aside from a uni- or bi-lateral tendinopathy of the patellar or Achilles tendon based on two clinical criteria: Tendon pain during physical activity and Tendon pain on local palpation.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2024-02-08 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Vessel density (all) | day 0 (the study is cross-sectional)
  Mean difference in blood vessel density detected by SURE imaging, between the healthy and tendinopathic group (across both patellar and Achilles).

SECONDARY OUTCOMES:
Repeatability (vessel density) | day 0 (the study is cross-sectional)
  Intraclass correlation of blood vessel density detected by SURE imaging in repeated ultrasound scans of the same tendon across all participants.

OTHER OUTCOMES:
Vessel density (PT/AT) | day 0 (the study is cross-sectional)
  Mean difference in blood vessel density detected by SURE imaging, between the healthy and tendinopathic group (within the patellar or Achilles individually).
Other quantifiable measures of microvasculature | day 0 (the study is cross-sectional)
  To-be-defined quantitative image analysis outcome of the microvasculature (due to the novelty of the method, the exact image analysis pipeline is not yet defined)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kjaer, PhD, Study Director — University Hospital Bispebjerg and Frederiksberg
Locations (1):
- Institute of Sports Medicine, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Due to the developmental nature of the study, the exact outcomes are currently poorly defined and the format in which they may be shared is therefore difficult to predict. We do intent to share individual participant data (IPD) in the form of to-be-defined image analysis outcomes as supplementary to relevant publications.